CLINICAL TRIAL: NCT02614703
Title: "Acetic Acid Chromoendoscopy in Barrett's Esophagus Surveillance is Superior to the Standardized Random Biopsy Protocol in Detecting Neoplasia: A Prospective Randomized Study"
Brief Title: "Acetic Acid Chromoendoscopy in Barrett's Esophagus Surveillance
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sample was under-powered
Sponsor: DHR Health Institute for Research and Development (Other)
Responsible Party: Principal Investigator, Ingrid Chacon, Gastroenterology Specialist, DHR Health Institute for Research and Development
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 0000001
Record Dates: First submitted 2015-07-30; First posted 2015-11-25 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Acetic Acid Chromoendoscopy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chromoendoscopy using Acetic Acid 2.5% (Experimental): Patient will have endoscopic examination of esophagus. Esophageal mucosa sprayed with 5cc solution of Acetic Acid 2.5% one time only. Esophageal mucosa examined again. Biopsies are obtained. Abnormal areas identified by Acetic Acid 2.5% will be submitted on separate containers for pathology review. If no abnormalities seen, random biopsies taken as per standard recommendations for Barrett's esophagus. Samples submitted for pathology review.
  Interventions: Drug: Chromoendoscopy using Acetic Acid 2.5%
- Standard random esophageal biopsies (Active Comparator): Patient will have endoscopic examination of the esophagus. Esophageal mucosa will not be sprayed with Acetic Acid 2.5%. Random biopsies taken as per standard recommendations for Barrett's esophagus. Samples submitted for pathology review.
  Interventions: Other: Standard random esophageal biopsies

INTERVENTIONS:
Drug: Chromoendoscopy using Acetic Acid 2.5% — Spraying esophageal mucosa during random biopsies for Barrett's esophagus
  Other Names: chromoendoscopy using ethanoic acid 2.5%
  Arms: Chromoendoscopy using Acetic Acid 2.5%
Other: Standard random esophageal biopsies — Random esophageal biopsies performed as per protocol
  Arms: Standard random esophageal biopsies

SUMMARY:
Neoplasia in Barrett's esophagus could be missed during routine random biopsies. We propose a study using chromoendoscopy with Acetic Acid to increase the yield of biopsies in detecting neoplasia.

DETAILED DESCRIPTION:
Neoplasia in Barrett's esophagus is often focal and can be missed by nontargeted biopsies alone. In recent years, various advanced endoscopic techniques have been utilized, but with varying success rates. Narrow-band imaging, trimodal imaging, spectral imaging and i-scan are technologies that are manufacturer dependent with limited varying success rates and have financial implications. At our institution, narrow band imaging is routinely utilized as a diagnostic tool for detecting Barrett's esophagus. Acetic acid is a commonly available dye that has been used in the detection of neoplasia in Barrett's esophagus.

This study is aimed to prove the effectiveness of acetic acid chromoendoscopy in our Barrett's esophagus surveillance population. The goal is to compare the neoplasia yield of acetic acid chromoendoscopy with that of standardized random biopsy protocol. The sensitivity and specificity for neoplasia detection by these two methods will also be analyzed.

Investigators plan to conduct this prospective randomized study for a period of one and a half years (beginning August 1, 2015, ending February 29, 2016). Based on data from 2014, we anticipate to enroll approximately 185 patients. All gastroenterologists (with privileges at Doctors Hospital at Renaissance) will participate in this study. Patients will be randomized to either acetic acid chromoendoscopy or current standard of care (standardized random biopsy protocol utilizing narrow band imaging). Random biopsies from both protocols and targeted biopsies (if identified) will be obtained and submitted to pathology department. These will be reviewed independently by two pathologists. Any discordant results will be reviewed by an outside expert pathologist. Statistical data analysis will be performed utilizing Datadesk XL software.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Previous diagnosis of Barrett's esophagus, confirmed by pathology.

Exclusion Criteria:

* Patients diagnosed with any level of dysplasia on previous esophageal biopsies.
* Patients who had esophageal therapy with Halo radiofrequency ablation in the past, or esophagectomy.
* History of allergy to Acetic Acid
* History of esophageal dysplasia or cancer
* Esophageal ulcerations
* Esophageal Candida
* Esophageal Varices
* Patients with active esophagitis
* Patients who cannot provide a valid consent
* Patients who are currently pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid M Chacon, MD, Principal Investigator — Doctor's Hospital at Renaissance
Locations (1):
- Doctors Hospital at Renaissance/Endoscopy Department, Edinburg, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual data available unless otherwise asked for safety reason.

REFERENCES:
- [Background] Longcroft-Wheaton G, Duku M, Mead R, Poller D, Bhandari P. Acetic acid spray is an effective tool for the endoscopic detection of neoplasia in patients with Barrett's esophagus. Clin Gastroenterol Hepatol. 2010 Oct;8(10):843-7. doi: 10.1016/j.cgh.2010.06.016. Epub 2010 Jun 30. PMID 20601133
- [Background] Tholoor S, Bhattacharyya R, Tsagkournis O, Longcroft-Wheaton G, Bhandari P. Acetic acid chromoendoscopy in Barrett's esophagus surveillance is superior to the standardized random biopsy protocol: results from a large cohort study (with video). Gastrointest Endosc. 2014 Sep;80(3):417-24. doi: 10.1016/j.gie.2014.01.041. Epub 2014 Apr 6. PMID 24713305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from our Barrett's esophageal Surveillance Program. The study took place in a South Texas Gastroenterology office. The first patient was enrolled 4-11-17. Study enrollment was stopped 7/30/18.
Pre-assignment Details: Patients were assigned an arm immediately after enrollment. There were no events within the enrollment and the actual procedure. The only reason patient could have been excluded was a no-show to the procedure appointment.
Groups:
- Standard Random Esophageal Biopsies: Patient will have endoscopic examination of the esophagus. Esophageal mucosa will not be sprayed with Acetic Acid 2.5%. Random biopsies taken as per standard recommendations for Barrett's esophagus. Samples submitted for pathology review.
  Standard random esophageal biopsies: Random esophageal biopsies performed one biopsy per quadrant, every 2cm of Barrett's mucosa ( also known as the Bethesta Protocol)
Period: Overall Study
Arm/Group | Chromoendoscopy Using Acetic Acid 2.5% | Standard Random Esophageal Biopsies
Started | 31 | 29
Completed | 24 | 28
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 7 | 1

BASELINE CHARACTERISTICS:
Population: Six patients randomized to the Acetic Acid arm, and four patients randomized to the standard random biopsies did not show to the test study by personal choice. Seven patients randomized to the Acetic Acid arm, and thirteen patients randomized to the Standard random esophageal biopsies did not have biopsy confirmed Barrett's esophagus.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chromoendoscopy Using Acetic Acid 2.5% | Standard Random Esophageal Biopsies | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 17 | 17 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 22 | 15 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 25 | 53
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
Number of participants with Long Segment Barrett's [Number; unit: participants] — Measurement of the length of Barrett's esophagus is performed during procedure. Length is reported in centimeters and is subjectively given by endoscopist performing procedure.
  Segments less than 3cm in maximal length are classified as short segment. Segments over 3cm in maximal length are classified as long segment.
  participants | 10 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Subjects With Neoplasia When Using Acetic Acid Chromoendoscopy Versus Standardized Random Biopsies.
Description: Spray of Acetic Acid into the esophageal mucosa during routine esophageal biopsies for Barrett's esophagus surveillance increases the yield of neoplasia.
Time Frame: 142 seconds
Population: Thirty-one (31) patients entered the preliminary data analysis. Of these 31 patients, twenty (20) were classified as SSBE, and eleven (11) patients as Long Segment BE (LSBE). These 31 patients were confirmed to have Barrett's esophagus via biopsy and were randomized (Acetic Acid n=20, Control n=11)
Measure: Number; unit: participants
Arm/Group | Chromoendoscopy Using Acetic Acid 2.5% | Standard Random Esophageal Biopsies
Number analyzed (Participants) | 20 | 11
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected upon completion of the procedure ( minutes to hours after the intervention/procedure). Patients were called 24 hours after the procedure and 48 hours after the procedure. Patients were evaluated at the office two weeks after the procedure.
Description: No adverse events were reported
Arm/Group | Chromoendoscopy Using Acetic Acid 2.5% | Standard Random Esophageal Biopsies
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT02614703/Prot_SAP_000.pdf